CLINICAL TRIAL: NCT02037516
Title: Does Residual Muscular Weakness Lead to an Increase in Respiratory Complications in Bariatric Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coastal Anesthesiology Consultants (Other)
Responsible Party: Principal Investigator, Patrick Ziemann-Gimmel, MD, Anesthesiologist, Principal Investigator, Coastal Anesthesiology Consultants
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAC
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Complication; Morbid Obesity
Keywords: residual muscle weakness, respiratory events
MeSH Terms: conditions — Obesity, Morbid | interventions — Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): qualitative monitoring of neuromuscular paralysis, standard treatment at this facility
  Interventions: Drug: Neostigmine; Device: Qualitative Monitor
- Study Group (Active Comparator): quantitative monitoring of neuromuscular paralysis as described in (Brull Murphy Anesth Analg 2010;111:129-40) Acceleromyography
  Interventions: Device: Accelomyography; Drug: Neostigmine

INTERVENTIONS:
Device: Accelomyography — quantitative measurement of the train-of-four with the TOF Watch to determine timing of administration of neostigmine and extubation To assure patient flow the time to reversal administration will be limited to approximately 30 minutes after achieving 4 twitches in qualitative monitoring
  Other Names: TOF watch
  Arms: Study Group
Drug: Neostigmine — Neostigmine is used to reverse the effects of neuromuscular blocking agents
Device: Qualitative Monitor — Qualitative (tactile or visual) assessment of residual neuromuscular paralysis
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if residual weakness after weight loss surgery leads to an increased risk of respiratory complications in the postoperative period.

DETAILED DESCRIPTION:
Patients interested in bariatric surgery would contact Dr. Marema or Dr. Koppman. Dr. Marema and Dr. Koppman will determine, if patients qualify for bariatric surgery. Patients will undergo a thorough preoperative workup. After optimization of all medical conditions patients would be scheduled for bariatric surgery. This is our current clinical practice.

One of the investigators would determine if a patient would qualify for the study. Then one of the investigators would approach the patients and explain the study in detail. Patients would be able to give informed consent or refuse to participate.

Patients refusing to participate in the study will need to sign a consent that data will be collect for internal quality control (IRB approval on file). The patients would be scheduled for bariatric surgery and be treated per our current clinical practice.

All patients would undergo a similar anesthetic. At the end of the procedure, before the NMBA reversal agent is given, the patients would be randomized to either the control or study group.

Intraoperative Anesthestic Management:

Patients receive sedative medication, typically midazolam 2-4mg iv. An infusion of dexmedetomidine will be started. Patients younger than 65 years will receive a loading dose of 1mcg/kg over 10 minutes. In patients older than 65 years 0.5 mcg/kg will be given as a loading dose. After administration of the loading dose an infusion will be continued throughout the duration of the surgery at a dose of 0.1-1mcg/kg/h. The infusion will be discontinued at the end of surgery. General anesthesia will be induced with a single dose of Lidocaine and Propofol with either Succinylcholine or Rocuronium given to provide intubating conditions. The patient's trachea will be intubated and mechanical ventilation started. General anesthesia will be maintained with an infusion of dexmedetomidine and propofol and titrated to the desired level of anesthesia. Ketamine will be administered as an adjunctive analgesic at a dose of 0.5 mg/kg. Neuromuscular blockade appropriate for surgical conditions will be provided by either the long acting neuromuscular blocking agents (NMBA), Rocuronium or Vecuronium, at the anesthesia providers discretion. At the conclusion of the operation the degree of NMB/paralysis will be assessed and a NMBA reversal administered (see detailed description below). Patients will be extubated after the end of surgery and transported to the PACU.

Monitoring of Neuro-Muscular Block (NMB or paralysis):

A signal is send from the brain to the muscle via an electrical impulse through a nerve. Electrical impulses can be applied externally to provoke muscle contraction. This technique is used to monitor the degree of paralysis induced by administration of NMBA.

NMBAs interrupt impulses or signals from the nerve to the muscle. External stimulation also does NOT lead to a muscle contraction in a paralyzed patient. Once the body metabolizes the NMBA the signal can travel again from the nerve to the muscle and provoke a muscle twitch. This recovery is gradual meaning that the initial twitches are weak and gradually get stronger. Also muscle fatigue faster with NMBA present (fade). This means that with similar, repetitive stimulation the twitch gets weaker. In anesthesia these attributes are examined to determine the degree of muscle relaxation and, or if at all, a dose of NMBA reversal can be given and what the appropriate dose should be.

There are two different ways of monitoring NMB: qualitative and quantitative.

Qualitative (current management) - Control Group:

The paralysis can be monitored tactile (feeling) or visual (seeing) to determine the twitch strength and the fade of repetitive stimulation. This determines the dose of reversal. After the reversal is given the anesthesia provider waits further to determine that the twitches are strong and there is no more fade. Then the patient will be extubated and transported to the PACU.

Quantitative (proposed management) - Study Group:

The paralysis would be monitored with a sensor (acceleromyography - AMG) that measures the twitch-strength after the ulnar nerve was stimulated (detailed explanation below). This objective data allows the anesthesia provider to titrate the NMBA reversal to best effect to assure adequate return to full muscle strength. Then the patient will be extubated and transported to the PACU.

AMG:

The technical term for the way of assessing the muscle contraction is called acceleromyography (AMG). AMG relies on 2 stimulating electrodes usually placed along the ulnar nerve at the wrist and a sensor that is placed in the groove between the thumb and the index finger; the sensor detects the acceleration of movement (bending) that is produced by the thumb in response to electrical stimulation of the ulnar nerve (TOF-Watch® SX Monitor). When the thumb contracts and accelerates the piezoelectric sensor, the degree of movement is sensed, and it is converted into electrical signals that are proportional to the force of thumb contraction. AMG can yield signals that can be measured and that can give an indication of the degree of neuromuscular block.

Randomization:

Patients will be randomized at the time when NMB can be reversed. Depending on the result the patient will be in the study or control group. Randomization will be done by a statistical software called R or an online web program called random.org.

Power analysis:

reduction from risk of a respiratory event in the postoperative period from 30% to 17.5% with an alpha of 0.05 and a power of 0.8 allocation approximately even in both groups (n1=n2) total sample size n=362, critical z=1.96, calculated by G Power 3

Data analysis:

primary Intention to treat analysis to reflect clinical reality, secondary analysis as per protocol

Definition of RE, adapted from Ziemann-Gimmel et. al. f1000research 2012 and Murphy et. al. Anesth Analg 2010;107(1):130-7

Protocol Changes:

Randomization occurs as described above at the time when the anesthesia provider feels "comfortable" based on the qualitative measurement of the TOF. If patient is randomized to the intervention group (quantitative measurement) reversal will be given based on the AMG (TOF Watch).

The change to the protocol:

1. If 30 minutes after the above time point no adequate AMG measurement is obtained reversal will be administered.
2. If after administration of reversal 30 minutes have elapsed and the AMG is less than 90% patients will be emerged from anesthesia.
3. administration of reversal in the intervention group will occur only after at least 4 twitches are measured consistently with the AMG. The previous suggested time-point suggested by the review article by Brull and Murphy where it can be given after 3 twitches seems to be to early and patients may not regain a TOF greater than 90%.

Dealing with missing TOF data:

If patients were randomized they will be analyzed in the according group (ITT). linear regression after log transformation will be done with the existing traces. There will be a best-/worst case scenario for sensitivity analysis. Missing values will be randomly sample and five scenarios will be analyzed to determine any impact (sensitivity analysis). (Imputation)

Also the best/worst case scenario will be analyzed:

best case: patients regain a TOF of 100% worst case: TOF is reduced by 5% from last measurement - it is physiologically unlikely that the TOF will be reduced to a greater extend over time.

ELIGIBILITY:
Inclusion Criteria:

- All patients scheduled for bariatric surgery at Flagler Hospital will be included after written and informed consent.

Exclusion Criteria:

- Patients will be excluded from the study if they don't consent to participate in the study. Patients allergic to any of the study medication will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Respiratory Events (RE) | 2 years
  Definition of RE, adapted from Ziemann-Gimmel et. al. f1000research 2012 and Murphy et. al. Anesth Analg 2010;107(1):130-7 Upper airway obstruction requiring an intervention; Hypoxemia despite 3 l/min NC requiring any intervention increasing FiO2 greater than 3 l/min NC tactile stimulation Signs of respiratory distress or impending ventilatory failure; Patient complaining of symptoms of respiratory or upper airway muscle weakness; w or w/o intervention Patient requiring reintubation in the PACU diagnosis of pneumonia on discharge or administration of antibiotics for suspected aspiration pneumonia unplaned application of CPAP/BiPAP unplanned ICU admission for respiratory reasons hypercarbic respiratory failure bag mask ventilation administration of "rescue" reversal after extubation for clinically suspected weakness prolonged intubation and ventilation in PACU and/or in ICU unplanned administration of breathing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ziemann-Gimmel, MD, Principal Investigator — Coastal Anesthesiology Consultants
Locations (1):
- Flagler Hospital, Saint Augustine, Florida, United States